CLINICAL TRIAL: NCT07272603
Title: Preliminary Clinical Study Evaluating the Therapeutic Response and Safety of Intravesical Perfusion With Plasma-Activated Saline Solution in Patients With Bladder Cancer
Brief Title: Bladder Perfusion of Plasma-Activated Saline for Bladder Cancer
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Benkang Shi, Head of Urology Department, Qilu Hospital of Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: bks05
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Bladder (Urothelial, Transitional Cell) Cancer
Keywords: bladder; cancer; Intravesical Perfusion; plasma
MeSH Terms: conditions — Neoplasms | interventions — Administration, Intravesical

STUDY DESIGN:
Intervention Model Description: This interventional study employs a single-arm, prospective, proof-of-concept model utilizing a within-subject control design, where each participant serves as their own baseline for comparison. The model leverages the pre-scheduled radical cystectomy as a definitive endpoint, allowing for a direct histological assessment of treatment effect. Efficacy is quantitatively measured by comparing pre- and post-treatment tumor volumes via MRI and analyzing the resected tissue for biomarkers of apoptosis, thereby providing a robust, paired analysis of the experimental intervention's biological impact within a short, controlled timeframe.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Plasma-Activated Saline Solution (PASS) Bladder Instillation (Experimental): This arm involves the intravesical instillation of the experimental intervention, Plasma-Activated Saline Solution (PASS), where 200 mL of the solution is administered into the bladder via a catheter every other day for 7 days, with a 1-hour dwell time, to evaluate its local efficacy in inducing tumor cell death and assess safety and tolerability.
  Interventions: Drug: Plasma-Activated Saline Solution (PASS) Bladder Instillation

INTERVENTIONS:
Drug: Plasma-Activated Saline Solution (PASS) Bladder Instillation — This intervention is distinguished by its unique mechanism of action, which utilizes physically-activated normal saline infused with reactive oxygen and nitrogen species (RONS) generated by non-thermal plasma, creating a potent yet transient cytotoxic solution that is administered locally.

SUMMARY:
This preliminary clinical study evaluates the safety and initial efficacy of a novel therapy called Plasma-Activated Saline Solution (PASS) for bladder cancer patients. The study involves a one-week course of PASS administered via bladder infusion in five pre-surgical patients, using imaging and pathology analyses to assess tumor shrinkage and cancer cell death, while closely monitoring for any adverse reactions to explore the therapy's future potential.

DETAILED DESCRIPTION:
This study is a prospective, proof-of-concept clinical trial investigating a novel local therapy for bladder cancer. The intervention involves the use of Plasma-Activated Saline Solution (PASS), a liquid infused with reactive oxygen and nitrogen species (RONS) created by exposing standard saline to cold atmospheric plasma. The goal is to leverage the potential of these activated substances to selectively target and kill cancer cells while minimizing damage to healthy bladder tissue.

The study will enroll a small cohort of five adult patients with confirmed bladder cancer who are already scheduled for a radical cystectomy (surgical removal of the bladder). This design allows for a direct assessment of the treatment's effect on the tumor within a short, controlled timeframe before surgery. Participants will receive intravesical (into the bladder) instillations of PASS every other day for one week, with each instillation retained for approximately one hour.

The primary objectives are twofold. First, to evaluate the treatment's efficacy, researchers will quantitatively measure the reduction in tumor volume using MRI scans conducted before and after the 7-day treatment period. Additionally, the surgically removed bladder tissue will be analyzed in the laboratory using immunohistochemistry to look for biological evidence of cancer cell death (apoptosis). Second, the study will rigorously assess safety and tolerability. This includes monitoring for severe, procedure-related adverse events and systematically tracking patient-reported symptoms like urinary pain and urgency using standardized diaries and scales.

As an initial exploratory investigation, this study is not designed to prove definitive clinical efficacy but to gather crucial first-in-human data on the biological activity and safety profile of PASS. The findings will determine whether this innovative approach warrants further development in larger clinical trials. The study will be conducted under strict ethical guidelines with close safety monitoring and full informed consent from all participants.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a pathological diagnosis of bladder cancer.
2. Patients scheduled for radical cystectomy, with at least one measurable tumor lesion ≥10 mm in diameter.
3. Age between 18 and 75 years.
4. Treatment-naïve patients who have not received any prior therapy for bladder cancer.

Exclusion Criteria:

1. Presence of severe comorbidities, including but not limited to cardiac disease, severe hepatic or renal insufficiency, uncontrolled hypertension, or diabetes.
2. Active urinary tract infection or a functional bladder capacity of less than 200 mL.
3. History of other malignancies.
4. Pregnancy or lactation.
5. Poor compliance, assessed as unlikely to complete the trial per protocol requirements.
6. Any other condition deemed by the investigator to make the patient unsuitable for study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Change in Tumor Size | Baseline (pre-treatment) and Day 7 (post-treatment).
  The reduction in tumor volume will be quantitatively assessed by comparing the product of the largest perpendicular diameters of the target tumor lesion measured on high-resolution magnetic resonance imaging (MRI) scans before and after the intervention.

SECONDARY OUTCOMES:
Proportion of Tumor Cells Undergoing Apoptosis | At the time of surgery (cystectomy), performed immediately following the 7-day intervention period.
  The biological effect on tumor cells will be evaluated through immunohistochemical analysis of biopsy specimens obtained during the post-treatment cystectomy, specifically measuring the percentage of tumor cells testing positive for TUNEL staining, which indicates programmed cell death (apoptosis).

CONTACTS AND LOCATIONS:
Overall Officials: benkang shi, Principal Investigator — Qilu Hospital of Shandong University

IPD SHARING:
Plan to Share IPD: No